CLINICAL TRIAL: NCT01682707
Title: Randomized Clinical Trials to Compare the Hemodynamic Response During Intubation Between Rigid Laryngoscopy and Track Light in Coronary Patients Undergoing CABG
Brief Title: Assessment of Hemodynamic Response During Intubation Between Rigid Laryngoscopy and Track Light in Coronary Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Marcello F Salgado Filho, MD, Master, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE-0021.0.185.000-09
Record Dates: First submitted 2010-04-01; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Disease Undergoing CABG
Keywords: intubation; coronary disease; hemodynamic response; anesthesia with tracheal intubation; assessment of hemodynamic response
MeSH Terms: conditions — Coronary Disease | interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laryngoscopy (Active Comparator): Laryngoscopy Track Light teaqueal intubation
  Interventions: Procedure: laryngoscopy
- Track Light (Active Comparator)
  Interventions: Procedure: track light

INTERVENTIONS:
Procedure: laryngoscopy — tracheal intubation with two different techniques, track light and laryngoscopy.
  Other Names: rigidy laryngoscopy,
  Arms: Laryngoscopy
Procedure: track light
  Arms: Track Light

SUMMARY:
Opioids provide greater patient comfort during intubation, but are not able to abolish completely the release adrenergic hormones during the laryngoscopy, which may cause undesirable hemodynamic changes.

In this study the investigators selected two techniques commonly used for intubation, laryngoscopy and track light, so the investigators can verify which intubation techniques provides less hemodynamic changes in coronary patients under standard anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* coronary disease ASA 2 e 3 using beta-blockers

Exclusion Criteria:

* emergency surgery arrythmia other antiarrythmic drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
hemodynamic response | patient prepare (baseline), 1min after induction, 5 min after induction, 1 min after intubation
  tracheal intubation with track light release less adrenergic hormones than laryngoscopy intubation

CONTACTS AND LOCATIONS:
Overall Officials: Marcello F Salgado filho, MD, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- National Institute of Cardiology / Ministry of Health, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Nishiyama T, Misawa K, Yokoyama T, Hanaoka K. Effects of combining midazolam and barbiturate on the response to tracheal intubation: changes in autonomic nervous system. J Clin Anesth. 2002 Aug;14(5):344-8. doi: 10.1016/s0952-8180(02)00370-7. PMID 12208438
- [Result] Nora FS, Klipel R, Ayala G, Oliveira Filho GR. [Remifentanil: does the infusion regimen make a difference in the prevention of hemodynamic responses to tracheal intubation?]. Rev Bras Anestesiol. 2007 Jun;57(3):247-60. doi: 10.1590/s0034-70942007000300003. Portuguese. PMID 19466360
- [Result] Almeida MC, Martins RS, Martins AL. [Tracheal intubation conditions at 60 seconds in children, adults and elderly patients.]. Rev Bras Anestesiol. 2004 Apr;54(2):204-11. doi: 10.1590/s0034-70942004000200007. Portuguese. PMID 19471727
- See also: Sociedade brasileira de Anestesiologia — http://www.sba.com.br
- See also: Related Info — http://www.inc.saude.gov.br
- See also: Related Info — http://www.scahq.org